CLINICAL TRIAL: NCT04880005
Title: Protocol for the Digital, Individualized, and Collaborative Treatment of Type 2 Diabetes in General Practice Based on Decision Aid (DICTA) - A Randomized Controlled Trial
Brief Title: Digital Individualized and Collaborative Treatment of T2D in General Practice Based on Decision Aid
Acronym: DICTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Steno Diabetes Center Odense (Other); Odense University Hospital (Other); Steno Diabetes Center Sjaelland (Other Government); Aalborg University (Other); Holbaek Sygehus (Other); Slagelse Sygehus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEA - DICTA
Record Dates: First submitted 2021-03-15; First posted 2021-05-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes type2
Keywords: diabetes type 2 management; digital behavioral coaching; lifestyle change; health behavior change; weight loss; interactive advice; participant engagement; quality of life
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The three core elements of the intervention are: 1) individualized data-driven recommendations to GPs on how to treat each individual T2D patient, as well as 2) individualized digital coaching of T2D patients, and 3) on-line presentation of patient registered outcomes (PRO) to GPs.
  Interventions: Behavioral: Clinical decision support; Behavioral: Digital Lifestyle Coaching; Behavioral: Integration to Standard Electronic Health Record
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Clinical decision support — Based on the phenotyping and algorithms developed by the hospital specialists at Odense University Hospital and Holbæk Hospital in collaboration with GPs, the individual GPs and their patients will receive individualized recommendations on lifestyle interventions and pharmacological treatments.
  The GPs will receive specific clinical decision support (CDS) recommendations on what drugs to prescribe to each patient based on the phenotyping in accordance with a clinical decision support tool (Cambio) and the updated guidelines at all times (Sparrow 2019). The treatment advice to the GPs will be adjusted annually based on treatment effect, re-phenotyping, and updated knowledge of the treatment of T2D. Furthermore, psychiatric, socioeconomic and/or cultural challenges and other determinants for frailty will be a part of the individualized intervention provided to patients by the GPs, again based on the specialist advice.
  Other Names: Individualized data-driven recommendations to GPs
  Arms: The intervention group
Behavioral: Digital Lifestyle Coaching — As part of DICTA, the patients are offered a personal health coach (dietician, nurse, occupational therapist, or physiotherapist) through the complex eHealth intervention (Liva). Patients will receive personalized empathic, relation driven coaching on healthy lifestyle on the individual patient's preferences (e.g. increased physical activity, healthier diet, weight loss, smoking cessation, personal goal setting, tailored information, peer to peer support), including optimal pharmacological treatment (Komkova 2019). The collaborative eHealth tool will give health coaches access to patient registered outcome measurements (PRO), information. This forms the basis of the individual coaching and is partly supported by artificial intelligence (AI) to improve the coaching by the health coaches (Holzinger 2016).
  Other Names: Individual digital coaching of T2D patients
  Arms: The intervention group
Behavioral: Integration to Standard Electronic Health Record — Data on physical activity, steps, diet goal fulfillment, smoking status etc., are being provided for GPs in a web-based solution integrated into the GPs' health record system. Integration with the GP system XMO (covering 52% of all Danish GPs) has been finalized.
  Other Names: Presentation of patient registered outcomes to GPs
  Arms: The intervention group

SUMMARY:
The purpose of this project is to improve life of patients with type 2 diabetes through an IT-supported lifestyle and treatment intervention.

The intervention is based on combining and adapting existing and effective elements into the IT system of the general practitioner. In this way we will integrate specialist supervised treatment in general practice, individual patient coaching, and improved information exchange and data mining.

The DICTA intervention consists of two integrated components: a patient-directed eHealth lifestyle coaching program delivered via the LIVA application, and a clinician-directed CDS tool embedded into the EPJ system.

1. eHealth lifestyle coaching: Individuals with T2D in the intervention group will receive individualized digital coaching from a health coach through the LIVA application. PROs are shared with GPs and health staff via the EPJ, enabling tailored, data-driven lifestyle support.
2. CDS: GPs receive real-time, individualized, algorithm-based pharmacological treatment recommendations for managing T2D, hypertension, and hypercholesterolemia, as appropriate.

This is expected to facilitate use, assure individually tailored solutions, optimize treatment effects, and strengthen patient engagement.

The study is a randomized controlled trial (RCT). It will include 400 patients with newly diagnosed type 2 diabetes. The patients will receive either treatment based on the intervention or usual care. After one year, we will assess quality of life and cardiovascular risk factors in both groups and evaluate if one group has improved management of their type 2 diabetes compared to the other.

If the intervention proves effective, implementation on a national scale is highly feasible, and the intervention could probably be adapted to other lifestyle-related chronic diseases in Denmark and in other countries.

DETAILED DESCRIPTION:
Background

A study from the UK showed that an intensive intervention comprising a total diet replacement, stepped food reintroduction and structured support for long-term weight loss maintenance resulted in long-term T2D remission for almost half of the patients (Lean et al., 2018).

In Denmark T2D is primarily managed in general practice, but despite intensive focus on T2D, many patients are not treated optimally, nor do they follow the recommendations for healthy lifestyle (Bo A et al, 2018). The Danish Center for Strategic Research in T2D (DD2) was initiated in 2010 with the overall aim of improving the quality of care for newly diagnosed T2D patients. The DD2 data comprises biological samples, as well clinical, lifestyle and quality of life data (Christensen et al, 2018). As of May 2019, DD2 holds samples from over 8,500 incident T2D patients. Based on the DD2 data, a model-intervention on individually tailored treatment of T2D was developed in 2013 and showed to be feasible in general practice (Stidsen et al, 2017).

Further researchers from the DICTA study group have found in a pilot study, a collaborative eHealth tool in a GP setting to induce weight loss among obese patients resulted in a 7 kg weight reduction, which was maintained over a 20-month period (Brandt et al., 2011) and a 5,4 kg weight loss for T2D men after 12 months (Haste et al, 2017). This collaborative eHealth tool(LIVA) has been updated and refined on the basis of input from extensive interviews with patients, healthcare professionals, and GPs (Brandt 2018a, Brandt 2018b and Brandt 2018c) and is in use in several Danish municipalities with promising results (Komkova 2019).

The DICTA project received support from Steno Collaboratory Grants 2018 and 2019 developing a web-based platform for patient registered outcome measurements and lifestyle coaching in collaboration with Liva Healthcare a/s, Cambio Healthcare Systems A/S and CGM A/S. This platform is now integrated in the electronic healthcare record systems used by the majority of Danish GPs (XMO, CGM). The intervention will provide novel, data-driven, individualized support to GPs, and individualized digital data-driven lifestyle support to their T2D patients supported by AI (machine learning) and timely accessible to the GPs when relevant.

Aim The study aims to determine whether this integrated digital approach can enhance patient engagement, support sustained behavior change, and improve health outcomes compared to usual care in general practice targeting management of T2D patients in a RCT.

Design and methods

Design:

The DICTA project is using a multi-method research approach including questionnaires, interviews, analysis of clinical outcome and health costs and all included in DICTA. This trial will recruit T2D patients in a GPs in the Region of Southern Denmark and Region of Zealand, and specialists from Odense University Hospital and Holbaek Hospital will electronically supervise the pharmacological treatment and specialized health coaches will offer online support for lifestyle changes. To ensure access to longitudinal data the investigators are aiming to enroll patients from GPs that also enroll their T2D patients in DD2. This will establish a comprehensive and strong inter-institutional and cross-sectional collaboration with the aim to improve care provided by the GPs and the quality of life for patients, based both on pharmacological and non-pharmacological treatments.

The intervention:

Based on the investigators previous research and subsequently developed IT programs and platforms, the investigators have implemented a complex intervention in collaboration with Liva Healthcare A/S, CGM and Cambio Healthcare Systems A/S. The two core elements of the intervention are:

1. Individualized supervised treatment Patients from DD2 who agree to participate have already been offered advanced phenotyping. Based on the phenotyping and algorithms developed by the hospital specialists at Odense University Hospital and Holbæk Hospital in collaboration with GPs. The GPs will receive specific clinical decision support recommendations on what drugs to prescribe to each patient based on the phenotyping in accordance with a clinical decision support tool (Cambio).
2. Individual digital coaching of T2D patients As part of DICTA, the patients are offered a personal health coach (dietician, nurse, occupational therapist, or physiotherapist) through the collaborative eHealth tool (Liva), and receive personalized empathic, relation driven coaching on healthy lifestyle on the individual patient's own terms (e.g. increased physical activity, healthier diet, weight loss, smoking cessation, personal goal setting, tailored information, peer to peer support), including optimal pharmacological treatment (Komkova, 2019). The collaborative eHealth tool will give health coaches access to patient registered outcome measurements (PROM) and support individual intervention goals. This forms the basis of the individual coaching and is partly supported by artificial intelligence (AI) to improve the coaching by the health coaches. As an example, health coaches are notified when patterns of usage is related to reduced success rates in weight loss. Presentation of patient registered outcomes to GPs Patient registered outcome measurements (PROM) on physical activity, steps, diet goal fulfillment, smoking status etc., are being provided for GPs in a web-based solution integrated into the GPs' health record system XMO, CGM (covering 52% of all Danish GPs).

Method In this RCT the investigators will test the effect of a combined individualized lifestyle and pharmacological treatment intervention package among newly diagnosed T2D patients in a GP setting. The investigators will recruit GPs from DD2 practices and invite new GPs to DD2 in Denmark. At each GP appointment, all patients newly diagnosed with T2D will be informed about the study in writing and orally, and those who agree to participate will after committing to informed consent via an online questionnaire be randomized 2:3 to either intervention or control group, after relevant time to consider if they want to participate, typically within one to two weeks. Inclusion will start May 3, 2021 and the investigators expect to have included all 400 patients by June 1, 2024. The intervention group receives one year of individualized treatment (the intervention) in addition to usual care, while the control group receives usual care in the first year and then both individualized treatment and usual care in the second year. This design enables analysis of the effect of the intervention after the first year August 31 2025. Both groups (intervention and control) will be seen by their GP at 3, 6, 9 and 12 months. No extra biological material will be collected in this study apart from what is collected as part of usual care and DD2.

Effect evaluation is displayed under outcome measures.

Sample size Based on our experience from the ongoing IDA trial the investigators expect that approximately 50% of the patients in the control group will meet the composite endpoint. With a minimal clinically relevant difference of 25%, at least 62.5% should meet the composite endpoint in the intervention group. With a power of 80% and a significance level of 5%, the investigators will need 200 patients in each group.

Statistical analysis The analyses will be performed by a statistician blinded to allocations. The primary analysis population will be the modified intention-to-treat population comprising those subjects with available data on the primary endpoint, i.e. those with completed 12-month follow-up. Per-protocol analyses will be predefined in the protocol and/or statistical analysis plan before any analyses are initiated. To enable the identification of the per-protocol population, major protocol deviations will be predefined in the protocol. To support future hypotheses, several ad-hoc exploratory analyses will also be performed. In general, categorical variables will be summarized as n (%), continuous variables as min-max, mean(sd), and median, Q1, Q3. All summaries will be by randomization group. Kaplan-Meier curves will be used to estimate survival functions related to time-to-event endpoints e.g. admissions stratified by group. Regression analyses, linear, logistic, and Cox proportional hazards will be used as appropriate. The type of analysis will depend on the endpoint in question. Before release of the data for analyses, a detailed statistical analysis plan will be written, reviewed, and approved.

Data Management

Through a collaboration with OPEN data will be collected using the online services provided in RedCap. In RedCap a project-specific and secure database can be developed for use in DICTA. This allows online and safe data sampling from all participating GP sites, and ensures a data handling process in concordance with current data protection legislation. Furthermore, RedCap supports automated integration between the eHealth solution and the GP-collected data, thus enabling merging of all data into one database. GP data will be laboratory results in accordance with the outcome descriptions as well as laboratory results, diagnose codes and medicine prescriptions of relevance for the clinical decision support tool developed in collaboration with Cambio. All statistics will be conducted via the service "OPEN analyze," placed on the same secure server as the project-specific OPEN database, or on the similarly protected research server at Statistics Denmark. A data management plan, including a protocol for access to and download of aggregated summaries and analysis results, will be available.

Dissemination of results

For the scientific dissemination, the investigators aim to publish in high-ranking scientific journals and present the data at scientific meetings, while at the same time pursuing the Science Europe principles on Open Access, ensuring the widest possible accessibility to the project outcomes.

Ethics

The overall assessment is that there are no risks of harm in project participation. Ethical permission will be obtained from the Danish Committee System on Health Research. Compliant to GDPR, written informed consent will be obtained from participants following an oral explanation of the project. Patient withdrawal from the study as well as the database can be done at any given time. All patient related data will be owned by SDCO. If ethical dilemmas should arise, experts at the involved institutions and ethical committees will be consulted. In case of disagreements, the PI decides about interpretation of data and on publication strategy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 in up to 10 years

Exclusion Criteria:

* Fails to complete the initial questionnaire
* No Internet access in own home through computer or smart phone
* Is pregnant or actively trying to get pregnant
* Has a serious or life-threatening disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in a binary indicator, composed by a composite endpoint of HbA1c, systolic blood pressure, low-density lipoprotein cholesterol, no smoking, and normal albuminuria | 12 months
  The primary outcome is the one-year change in estimated ten-year cardiovascular risk assessed by SCORE2-Diabetes calculated from age, smoking status, systolic blood pres-sure, total and high-density lipoprotein cholesterol, age at diabetes diagnosis, HbA1c, and eGFR. As we will be focusing on one-year changes in SCORE2-Diabetes, we do not consider it a problem that SCORE2-Diabetes does not include prevalent cardiovascular disease in the risk calculation as this variable will be constant over the one-year period on almost all of the patients.

SECONDARY OUTCOMES:
Change in HbA1c | 12 months
  Measured in mmol/mole as the number of persons with HbA1c less than 53 mmol/mole
Numbers change in level of use of hypertension, hypercholesterolemic and glucose-lowering drugs | 12 months
  Number of patients change in medication in accordance with the following guideline:
  Increased:
  1. increased dosage of known drug
  2. adding extra drug
  No change
  1. same drug before and after
  2. shift to another drug i.e. metformin to SGLT2 inhibitor or Victoza to Ozempic
  Reduced:
  1. reduced dosage of known drug
  2. reducing number of drugs
Change in quality of life measured by European Quality of life - 5 Dimensions - 5 level (EQ-5D-5L) | 12 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in weight | 12 months
  Measured in kilograms
Change in abdominal circumference to hip circumference | 12 months
  Ratio measured in centimeters to centimeters
Change in physical activity measured through AX3 | 12 months
  Measured in minutes of activity
Change in systolic blood pressure | 12 months
  Measured in mmHg as the number of persons with less than 140 mmHg
Change in low-density lipoprotein cholesterol | 12 months
  Measured in mmol/L and mg/dl as the number of persons with less than 2.5mmol/l or 97mg/dl
Change in number of patients not smoking, | 12 months
  Measured as the number of patients who do not smoke
Change in level of albuminuria | 12 months
  Measured in urine albumin/creatinine ratio * 10-3 as as the number of persons with less than 30 *10-3
Change in HbA1c | 12 months
  Measured in mmol/mole as the number of persons with HbA1c less than 48 mmol/mole
Change in quality of life measured by European Quality of life - EQ VAS | 12 months
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale (0-100), where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Jens H Søndergaard, Principal Investigator — University of Southern Denmark
Locations (1):
- Research Unit for General Practice, Department for Public Health, University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be made accessible after end of study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will become available when published starting july of 2022 and to be held accessible until January 2030
Access Criteria: Accessible partly on the website and partly upon request to the PI
URL: http://www.dicta.dk

REFERENCES:
- [Background] Bo A, Thomsen RW, Nielsen JS, Nicolaisen SK, Beck-Nielsen H, Rungby J, Sorensen HT, Hansen TK, Sondergaard J, Friborg S, Lauritzen T, Maindal HT. Early-onset type 2 diabetes: Age gradient in clinical and behavioural risk factors in 5115 persons with newly diagnosed type 2 diabetes-Results from the DD2 study. Diabetes Metab Res Rev. 2018 Mar;34(3). doi: 10.1002/dmrr.2968. Epub 2017 Dec 21. PMID 29172021
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132
- [Background] Christensen DH, Nicolaisen SK, Berencsi K, Beck-Nielsen H, Rungby J, Friborg S, Brandslund I, Christiansen JS, Vaag A, Sorensen HT, Nielsen JS, Thomsen RW. Danish Centre for Strategic Research in Type 2 Diabetes (DD2) project cohort of newly diagnosed patients with type 2 diabetes: a cohort profile. BMJ Open. 2018 Apr 7;8(4):e017273. doi: 10.1136/bmjopen-2017-017273. PMID 29627803
- [Background] Stidsen JV, Nielsen JS, Henriksen JE, Friborg SG, Thomsen RW, Olesen TB, Olsen MH, Beck-Nielsen H. Protocol for the specialist supervised individualised multifactorial treatment of new clinically diagnosed type 2 diabetes in general practice (IDA): a prospective controlled multicentre open-label intervention study. BMJ Open. 2017 Dec 10;7(12):e017493. doi: 10.1136/bmjopen-2017-017493. PMID 29229652
- [Background] Brandt V, Brandt CJ, Glintborg D, Arendal C, Toubro S, Brandt K Sustained Weight Loss during 20 Months using a Personalized Interactive Internet Based Dietician Advice Program in a General Practice Setting, International Journal on Advances in Life Sciences, vol 3 no 1 & 2, year 2011,
- [Background] Haste A, Adamson AJ, McColl E, Araujo-Soares V, Bell R. Web-Based Weight Loss Intervention for Men With Type 2 Diabetes: Pilot Randomized Controlled Trial. JMIR Diabetes. 2017 Jul 7;2(2):e14. doi: 10.2196/diabetes.7430. PMID 30291100
- [Background] Brandt CJ, Clemensen J, Nielsen JB, Sondergaard J. Drivers for successful long-term lifestyle change, the role of e-health: a qualitative interview study. BMJ Open. 2018 Mar 12;8(3):e017466. doi: 10.1136/bmjopen-2017-017466. PMID 29530904
- [Background] Brandt CJ, Sogaard GI, Clemensen J, Sndergaard J, Nielsen JB. General Practitioners' Perspective on eHealth and Lifestyle Change: Qualitative Interview Study. JMIR Mhealth Uhealth. 2018 Apr 17;6(4):e88. doi: 10.2196/mhealth.8988. PMID 29666045
- [Background] Brandt CJ, Sogaard GI, Clemensen J, Sondergaard J, Nielsen JB. Determinants of Successful eHealth Coaching for Consumer Lifestyle Changes: Qualitative Interview Study Among Health Care Professionals. J Med Internet Res. 2018 Jul 5;20(7):e237. doi: 10.2196/jmir.9791. PMID 29980496
- [Background] Komkova A, Brandt CJ, Hansen Pedersen D, Emneus M, Sortso C. Electronic Health Lifestyle Coaching Among Diabetes Patients in a Real-Life Municipality Setting: Observational Study. JMIR Diabetes. 2019 Mar 12;4(1):e12140. doi: 10.2196/12140. PMID 30860486